CLINICAL TRIAL: NCT02833077
Title: A Multicenter, Single-blind, Randomized, Controlled Study of the Safety and Effectiveness of JUVÉDERM VOLUMA® XC Injectable Gel for Chin Augmentation
Brief Title: A Safety and Effectiveness Study of JUVÉDERM VOLUMA® XC Injectable Gel for Chin Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Voluma-006
Record Dates: First submitted 2016-07-12; First posted 2016-07-14 (Estimated); Results first posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Chin Retrusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- JUVÉDERM VOLUMA® XC (Experimental): JUVÉDERM VOLUMA® XC was injected into the chin at a volume determined by the investigator on Day 0. Participants were eligible to receive touch-up treatment 30 days later, if applicable. The maximum total volume administered was up to 4 milliliters (mL) for both treatments combined.
  Interventions: Device: JUVÉDERM VOLUMA® XC
- No Treatment then JUVÉDERM VOLUMA® XC (Other): No treatment for 6 months followed by optional treatment with JUVÉDERM VOLUMA® XC injected into the chin at a volume determined by the investigator on Month 6. Participants were eligible to receive touch-up treatment 30 days later, if applicable. The maximum total volume administered was up to 4 mL for both treatments combined.
  Interventions: Device: JUVÉDERM VOLUMA® XC

INTERVENTIONS:
Device: JUVÉDERM VOLUMA® XC — JUVÉDERM VOLUMA® XC was injected into the chin at a volume determined by the investigator. The maximum total volume administered was up to 4 mL.

SUMMARY:
This is a safety and effectiveness study of JUVÉDERM VOLUMA XC injectable gel for chin augmentation to correct volume deficit in chin retrusion.

ELIGIBILITY:
Inclusion Criteria:

* Chin retrusion
* In good general health

Exclusion Criteria:

* Permanent facial implants on the face and/or neck
* Received fat injections below the nose
* Tattoos, piercings, beard, mustache, and/or scars on the face below the nose
* Received semi-permanent dermal fillers in the chin or jaw line in the last 3 years
* Undergone dermal filler injections or had any surgery in the chin or jaw area in the last 2 years
* Received dermal filler injections in the lips or in the mouth area in the last 12 months
* Undergone mesotherapy or cosmetic treatment (e.g., laser, photomodulation, intense pulsed light, radio frequency, dermabrasion, moderate or greater depth chemical peel, liposuction, lipolysis, or other ablative procedures) anywhere in the face or neck in the last 6 months
* Received botulinum toxin treatment below the nose in the last 6 months

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2016-06-28 (Actual); Primary Completion 2018-02-06 (Actual); Study Completion 2018-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Schumacher, Study Director — Allergan
Locations (14):
- United States (14):
  - Dermatology Cosmetic Laser Medical Associates of La Jolla, Inc., San Diego, California
  - Skin Research Institute, Coral Gables, Florida
  - Baumann Cosmetic and Res. Institute, Miami Beach, Florida
  - Research Institute of the Southeast, West Palm Beach, Florida
  - DeNova Research, Chicago, Illinois
  - Callender Dermatology and Cosmetic Center, Glenn Dale, Maryland
  - SkinCare Physicians of Chestnut Hill, Chestnut Hill, Massachusetts
  - St Louis University Medical Center Dept. of Dermatology, St Louis, Missouri
  - Image Dermatology, PC, Montclair, New Jersey
  - Williams Plastic Surgery Specialists, Latham, New York
  - The Center for Dermatology, Cosmetics, & Laser Surgery, Mount Kisco, New York
  - Dermatology & Laser Center of Charleston Center for Clinical Research, Charleston, South Carolina
  - Nashville Centre for Laser and Facial Surgery, Nashville, Tennessee
  - Premier Clinical Research; Spokane Dermatology Clinic, Spokane, Washington

REFERENCES:
- [Derived] Beer K, Kaufman-Janette J, Bank D, Biesman B, Dayan S, Kim W, Chawla S, Schumacher A. Safe and Effective Chin Augmentation With the Hyaluronic Acid Injectable Filler, VYC-20L. Dermatol Surg. 2021 Jan 1;47(1):80-85. doi: 10.1097/DSS.0000000000002795. PMID 33347003
- See also: More Information — http://www.allerganclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 221 participants were enrolled in the study, with enrollment defined as signing the informed consent form. A total of 29 enrolled participants were screen failures (did not meet eligibility criteria). Thus, a total of 192 participants were randomized.
Period: Overall Study
Arm/Group | JUVÉDERM VOLUMA® XC | No Treatment Then JUVÉDERM VOLUMA® XC
Started | 144 | 48
Participants Treated | 144 | 38
Completed | 127 | 40 (Includes participants who completed the study but did not receive the optional treatment.)
Not Completed | 17 | 8
Not completed — Adverse Event | 1 | 2
Not completed — Lost to Follow-up | 10 | 1
Not completed — Personal Reasons | 6 | 4
Not completed — Protocol Deviation | 0 | 1

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-Treat (mITT) Population included all participants randomized to the treatment group who received at least 1 study treatment or all participants randomized to the control group.
Groups:
- JUVÉDERM VOLUMA® XC: JUVÉDERM VOLUMA® XC was injected into the chin at a volume determined by the investigator on Day 0. Participants were eligible to receive touch-up treatment 30 days later, if applicable. The maximum total volume administered was up to 4 mL for both treatments combined.
- Total: Total of all reporting groups
Arm/Group | JUVÉDERM VOLUMA® XC | No Treatment Then JUVÉDERM VOLUMA® XC | Total
Number analyzed (Participants) | 144 | 48 | 192
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (13.4) | 48.9 (14.3) | 49.8 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129 | 41 | 170
  Male | 15 | 7 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 6 | 33
  Not Hispanic or Latino | 117 | 42 | 159
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 23 | 6 | 29
  White | 116 | 41 | 157
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  North America | 144 | 48 | 192

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a ≥ 1-point Improvement (Decrease) on the Allergan Chin Retrusion Scale (ACSR) Score
Description: The evaluating investigator assessed the participant's chin retrusion based on 2-dimensional (2D) renderings of 3-dimensional (3D) images using the validated 5-point photonumeric ACRS where: 0= None (no chin retrusion) to 4=Extreme (extreme chin retrusion).
Time Frame: Baseline (up to 30 days prior to randomization) to Month 6
Population: The mITT population included all participants randomized to the treatment group who received at least 1 study treatment or all participants randomized to the control group. Overall number of participants analyzed were the participants with analysis values at both Baseline and Post-baseline during the specified time period.
Measure: Number; unit: percentage of participants
Arm/Group | JUVÉDERM VOLUMA® XC | No Treatment Then JUVÉDERM VOLUMA® XC
Number analyzed (Participants) | 126 | 40
percentage of participants | 56.3 | 27.5
Statistical Analysis 1: Comparison: JUVÉDERM VOLUMA® XC vs No Treatment Then JUVÉDERM VOLUMA® XC; Superiority of treatment group was established if responder rate at month 6 was statistically greater than that for the control group at month 6 and the observed responder rate at month 6 for the treatment group was greater than 50%; Test type: Superiority; p = 0.0019, Fisher's exact test — If the 2-sided p-value is < 0.05, the responder rate is greater for treatment than for control group, and point estimate of the responder rater for treatment group is greater than 50%, then treatment will be considered superior to control group; Responder Rate Difference = 28.85, 95% CI 2-sided [11.16 to 45.60]

2. Secondary Outcome: Change From Baseline in Overall Scores of the Satisfaction With Chin Module of the FACE-Q Questionnaire
Description: The participant answered 10 question on the chin module of the FACE-Q about their satisfaction with their chin using a 4-point scale where: 1=Very Dissatisfied, 2=Somewhat Dissatisfied, 3=Somewhat Satisfied and 4=Very Satisfied. The total score was transformed to a score of 0 (worse) to 100 (best). A positive change from Baseline indicates improvement.
Time Frame: Baseline (up to 30 days prior to randomization) to Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | JUVÉDERM VOLUMA® XC | No Treatment Then JUVÉDERM VOLUMA® XC
Number analyzed (Participants) | 126 | 40
score on a scale
  Baseline | 35.7 (17.7) | 35.3 (14.9)
  Change from Baseline to Month 6 | 35.6 (23.2) | -3.3 (11.5)
Statistical Analysis 1: Comparison: JUVÉDERM VOLUMA® XC; Test type: Other; p < .0001, Two sided paired t-test — P-value is based on a 2-sided paired t-test at the 5% level to demonstrate that the mean overall satisfaction score at month 6 visit is statistically greater than that at the baseline for the treatment group

3. Secondary Outcome: Percentage of Participants Improved or Much Improved on the 5-Point Global Aesthetic Improvement Scale (GAIS) for the Chin Area As Assessed by the Evaluating Investigator
Description: The evaluating investigator assessed the participant's chin area using the GAIS where: 2=Much Improved, 1=Improved, 0=No change, -1=Worse and -2=Much Worse.
Time Frame: Baseline (up to 30 days prior to randomization) to Month 6
Population: The mITT population included all participants randomized to the treatment group who received at least 1 study treatment or all participants randomized to the control group. Overall number analyzed is the number of participants with data available for analyses.
Measure: Number; unit: percentage of participants
Arm/Group | JUVÉDERM VOLUMA® XC | No Treatment Then JUVÉDERM VOLUMA® XC
Number analyzed (Participants) | 125 | 41
percentage of participants | 91.2 | 19.5

4. Secondary Outcome: Percentage of Participants Improved or Much Improved on the 5-Point GAIS for the Chin Area As Assessed by the Participants
Description: The participants who received JUVÉDERM VOLUMA® XC, assessed their chin area using the GAIS where: 2=Much Improved, 1=Improved, 0=No change, -1=Worse and -2=Much Worse.
Time Frame: Baseline (up to 30 days prior to randomization) to Month 6
Population: Participants in the mITT population who were randomized to the treatment group and received at least 1 study treatment with available data were included in the analyses.
Measure: Number; unit: percentage of participants
Arm/Group | JUVÉDERM VOLUMA® XC
Number analyzed (Participants) | 126
percentage of participants | 87.3

ADVERSE EVENTS:
Time Frame: JUVÉDERM VOLUMA® XC: Up to 12 months following treatment. No Treatment then JUVÉDERM VOLUMA® XC: Up to 6 months during No Treatment; Up to 6 months following treatment (Up to Month 12)
Description: Safety population included all participants randomized to the treatment group who received at least 1 study device treatment or all participants randomized to the control group.
Groups:
- No Treatment: Participants who received no treatment for the first 6 months.
- JUVÉDERM VOLUMA® XC After No Treatment: Participants who received optional treatment with JUVÉDERM VOLUMA® XC injected into the chin at a volume determined by the investigator on Month 6 after no treatment for 6 months. Participants were eligible to receive touch-up treatment 30 days later, if applicable. The maximum total volume administered was up to 4 mL for both treatments combined.
Arm/Group | JUVÉDERM VOLUMA® XC | No Treatment | JUVÉDERM VOLUMA® XC After No Treatment
All-Cause Mortality (participants affected / at risk) | 0/144 | 0/48 | 0/38
Serious Adverse Events (participants affected / at risk) | 10/144 | 4/48 | 1/38
Other Adverse Events (participants affected / at risk) | 0/144 | 0/48 | 0/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | JUVÉDERM VOLUMA® XC (N=144) | No Treatment (N=48) | JUVÉDERM VOLUMA® XC After No Treatment (N=38)
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Injection site cellulitis (Infections and infestations) | 1 | 0 | 0
Injection site inflammation (General disorders) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Invasive papillary breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Breast cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-02-28): https://cdn.clinicaltrials.gov/large-docs/77/NCT02833077/SAP_000.pdf
  • Study Protocol (2017-03-01): https://cdn.clinicaltrials.gov/large-docs/77/NCT02833077/Prot_001.pdf